CLINICAL TRIAL: NCT04983550
Title: A Multicenter, Randomized, Controlled, Open-label, Phase II Study to Evaluate the Efficacy and Safety of SG001 in Combination With PLD in Patients With Platinum-resistant Relapsed Epithelial Ovarian Cancer
Brief Title: Efficacy and Safety of SG001 Combined With PLD in Patients With Platinum-resistant Relapsed EOC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYSA1802-CSP-003
Record Dates: First submitted 2021-07-16; First posted 2021-07-30 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Epithelial Ovarian Cancer; Fallopian Tube Cancer; Peritoneal Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — 1-dodecylpyridoxal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: SG001 + doxorubicin hydrochloride liposome injection (Experimental): Two-thirds of the patients will be randomly assigned to group A to receive SG001 240 mg, IV, every 2 weeks (1 cycle every 4 weeks), and doxorubicin hydrochloride liposome injection 40 mg/m^2, IV, every 4 weeks (1 cycle).
  Interventions: Drug: SG001; Drug: Doxorubicin hydrochloride liposome injection
- Group B: doxorubicin hydrochloride liposome injection (Active Comparator): One-third of the patients will be randomly assigned to group B to receive doxorubicin hydrochloride liposome injection 40 mg/m^2, IV, every 4 weeks (1 cycle).
  Interventions: Drug: Doxorubicin hydrochloride liposome injection

INTERVENTIONS:
Drug: SG001 — Recombinant Anti-PD-1 Fully Human Monoclonal Antibody Injection, 240 mg q2w
  Other Names: Recombinant Anti-PD-1 Fully Human Monoclonal Antibody Injection
  Arms: Group A: SG001 + doxorubicin hydrochloride liposome injection
Drug: Doxorubicin hydrochloride liposome injection — Doxorubicin hydrochloride liposome injection 40mg/m ^2 q4w
  Other Names: PLD

SUMMARY:
This study is a multicenter, randomized, controlled, open-label, phase II study to evaluate the efficacy and safety of SG001 in combination with doxorubicin hydrochloride liposome injection in patients with platinum-resistant relapsed epithelial ovarian cancer.

DETAILED DESCRIPTION:
This is a multicenter, randomized, controlled, open-label, phase II clinical study to evaluate the efficacy and safety of SG001 in combination with doxorubicin hydrochloride liposome injection in patients with platinum-resistant relapsed intermediate to advanced epithelial ovarian cancer, and to provide a basis for recommending the SG001 combination dosing regimen for subsequent studies. This study will enroll patients with histologically or cytologically confirmed epithelial ovarian, fallopian tube, or peritoneal cancer, FIGO stage II-IV, platinum-resistant relapse (defined as disease progression within 6 months after the last platinum-containing chemotherapy) and non-platinum refractory (defined as disease progression within 4 weeks after the first platinum-containing chemotherapy) with up to three prior lines of platinum-containing systemic chemotherapy, up to two lines of platinum-free systemic chemotherapy, and at least one measurable tumor lesion (according to RECIST 1.1).

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 18-75 (inclusive) years old (based on the day of signing the informed consent).
2. Histologically or cytologically confirmed epithelial ovarian, fallopian tube, or peritoneal, FIGO stage II-IV (per FIGO 2014).
3. Patients with platinum-resistant relapse (defined as disease progression within 6 months after the last platinum-containing chemotherapy) and non-platinum refractory (defined as disease progression within 4 weeks after the first platinum-containing chemotherapy). Previously received up to three lines of platinum-containing system chemotherapy and up to two lines of platinum-free system chemotherapy.
4. Patients must provide sufficient qualified FFPE tumor tissue specimens or sections for PD-L1 detection.
5. At least one measurable lesion per RECIST 1.1 at baseline. Measurable lesions should not have received local treatment such as radiotherapy (lesions located within previous radiotherapy areas may also be selected as a target lesion if progression is confirmed).
6. Eastern Cooperative Oncology Group (ECOG) physical status score: 0 or 1.
7. Life expectancy ≥3 months.
8. Vital organ function meets the following requirements (no blood transfusion, no use of hematopoietic stimulating factor, and no use of medication to correct blood cell count within 14 days prior to first administration):

   A) Absolute neutrophil count (ANC) ≥ 1.5×10^9/L; B) Platelet count (PLT) ≥ 75×10^9/L; C) Hemoglobin (HGB) ≥ 9 g/dL; D) Serum creatinine Cr ≤ 1.5×ULN or creatinine clearance Ccr ≥ 50 mL/min; E) Total bilirubin (TBil) ≤ 1.5×ULN (3×ULN for patients with Gilbert's syndrome); F) Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×ULN (≤ 5×ULN for patients with liver metastasis); G) Activated partial thromboplastin time (APTT) and international standardized ratio (INR) ≤ 1.5×ULN (no correction with anticoagulants or other drug affecting coagulation function within 14 days before the first administration, except long-term anticoagulant therapy is needed.).
9. Toxic and side effects caused by previous anti-tumor therapy should be restored to ≤1 grade (CTCAE 5.0) (except residual alopecia and fatigue) before enrollment.
10. Patients are required to give informed consent to this study and voluntarily sign a written informed consent prior to the study.

Exclusion Criteria:

1. A history of severe allergic reaction and uncontrolled allergic asthma to monoclonal antibody preparations.
2. Untreated known CNS metastases, or treated CNS metastases but still with symptoms (except for residual signs or symptoms related to CNS treatment, and those with stable or improved neurological symptoms for at least 2 weeks prior to screening can be enrolled).
3. Patients with a history of primary immunodeficiency.
4. Patients with an active autoimmune disease or a history of autoimmune disease, but with well-controlled type Ⅰ diabetes, well-controlled hypothyroidism requiring only hormone replacement therapy, skin conditions that do not require general treatment (such as vitiligo, psoriasis, or alopecia), or patients whose disease is not expected to recur in the absence of external triggers, will be screened for further enrollment.
5. Baseline cardiac ejection fraction is less than 50% or the lower limit of normal; history of clinically significant prolonged QTc interval (> 450 ms in male, > 470 ms in female); cardiac lesions caused by previous use of anthracyclines; serious cardiovascular disease, such as New York Heart Association (NYHA) grade 2 or higher heart failure, previous myocardial infarction within 3 months, poorly controlled arrhythmias, or unstable angina.
6. Severe arterial/venous thrombosis events (such as transient ischemic attack, cerebral haemorrhage, cerebral infarction, deep venous thrombosis, pulmonary embolism, etc.) within 3 months prior to screening.
7. Previous interstitial lung disease (except local interstitial pneumonia induced by radiotherapy), non-infectious pneumonia requiring glucocorticoid therapy.
8. Have received any other antibodies/drugs that act on T cell co-stimulation or checkpoint pathways (including PD-1, PD-L1, PD-L2, CTLA-4, OX40, C137 inhibitors, etc.).
9. Patients with immune related AE CTCAE 5.0 grade score ≥ 3 after receiving immunotherapy.
10. Major surgery or radical radiotherapy within 28 days prior to the first administration, or palliative radiotherapy within 14 days prior to the first administration, or radiation agents (strontium, samarium, etc.) within 56 days prior to the first administration.
11. Those who have received systemic antitumor therapy, including but not limited to chemotherapy, immunotherapy, macromolecular targeted therapy, or biotherapy (tumor vaccines, cytokines, or growth factors for cancer control) within 28 days before the first administration of the drug; small molecule targeting and oral fluorouracil-based therapy within 14 days (or 5 half-lives, whichever is longer) prior to first administration; those who had received mitomycin C and nitrosourea within 6 weeks prior to initial administration.
12. Those who received live attenuated vaccine within 28 days before the first administration or who planned to receive it during the study period.
13. Any active infection that requires systemic treatment by intravenous drip within 28 days prior to first administration.
14. Those who have received treatment within 14 days prior to the first dose with a proprietary Chinese medicine that has a clear antitumor-related function in the NMPA-approved drug specification or a Chinese herbal medicine that is clearly documented in the medical record for antitumor purposes.
15. Patients who have received whole or component blood transfusion within 14 days prior to initial administration.
16. Glucocorticoids (prednisone >10 mg/day or equivalent of another similar drug) or other immunosuppressive therapy for a condition within 14 days prior to first administration.
17. Participation in other clinical trials and use of the investigational drug within 28 days prior to the first administration (counting from the date of the last treatment in the previous clinical study) (with the exception of the overall survival follow-up period in one study).
18. Positive for human immunodeficiency virus (HIV-Ab) and treponema pallidum antibody (TP-Ab) antibodies; positive for hepatitis B virus surface antigen (HBsAg) and/or hepatitis B core antibody (HBcAb), with HBV quantitative detection value > upper limit of normal value; positive for hepatitis C antibody (HCV-Ab), with hepatitis C virus RNA quantification > upper limit of normal value.
19. History of active tuberculosis.
20. Pregnant or breastfeeding women.
21. Known suffered from other malignant tumors that have progressed or require treatment within 5 years prior to screening (except for well-treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer or cured carcinoma in situ, such as breast carcinoma in situ, etc.).
22. Other circumstances that may increase the risk associated with the study medication, or interfere with the interpretation of the study results, or affect the compliance of the study, etc. may not be suitable for participation in the study as determined by the investigator.
23. Previous use of doxorubicin liposomes.
24. Previous use of other anthracycline/anthraquinone drugs (including non-doxorubicin liposomes) with a converted cumulative dose equivalent to doxorubicin ≥300 mg/m^2, or previous use of anthracyclines causing cardiac disease.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
1. Objective response rate (ORR, assessed by investigators according to RECIST 1.1 criteria) | From date of first drug administration until the first documented progression of disease, patient withdrawal, lose to follow-up, death, initiating a subsequent cancer therapy, or study completion or termination, whichever occurs earliest.
  ORR is defined as the proportion of all patients with a best evaluation of complete response or partial response (according to RECIST version 1.1 criteria), from the date of administration to the date of patients' withdrawal or study completion or termination.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | From date of first drug administration until the first documented progression of disease, patient withdrawal, lose to follow-up, death, initiating a subsequent cancer therapy, or study completion or termination, whichever occurs earliest,up to 3 years.
  PFS measured from the date of administration to the date of investigator firstly assessed disease progression (according to RECIST version 1.1 criteria) or death from any cause (in the absence of progression).
Disease control rate (DCR) | From date of first drug administration until the first documented progression of disease, patient withdrawal, lose to follow-up, death, initiating a subsequent cancer therapy, or study completion or termination, whichever occurs earliest,up to 2 years.
  DCR is defined as the proportion of all patients with best a evaluation of complete response or partial response or stable disease (according to RECIST version 1.1 criteria) from the date of administration to the date of patients' withdrawal or study completion or termination.
Overall survival (OS) | From date of first drug administration until the first documented progression of disease, patient withdrawal, lose to follow-up, death, initiating a subsequent cancer therapy, or study completion or termination, whichever occurs earliest,up to 3years..
  OS measured from the date of administration to the date of death from any cause.
Treatment emergent adverse event (TEAEs) | From the date of signing Informed Consent Form (ICF) up to 28 days following the last dose of study drug, immune related adverse events will be recorded until 90 days after the last dose.
  Amount, severity, and duration of TEAEs will be evaluated according to NCI-CTCAE V5.0.